CLINICAL TRIAL: NCT06307015
Title: De-escalation of Radiation Dose in HPV-associated Oropharyngeal Squamous Cell Carcinoma Utilising FMISO PET and Magnetic Resonance Imaging as Non-Invasive Biomarkers of Hypoxia (DE-RADIATE)
Brief Title: De-escalation of Radiation Dose in HPV-associated OPC Utilising FMISO PET (DE-RADIATE)
Acronym: DE-RADIATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Anna Lawless, Radiation Oncology Fellow & Principal Investigator, Royal North Shore Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/ETH02441
Record Dates: First submitted 2024-03-01; First posted 2024-03-12 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-04

CONDITIONS: HPV Positive Oropharyngeal Squamous Cell Carcinoma
Keywords: Radiation therapy; De-escalation; FMISO PET; Hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (Active Comparator): Standard of care treatment for patients undergoing definitive chemoradiation for oropharyngeal squamous cell carcinoma
  Interventions: Radiation: Standard of care
- De-escalation (Experimental): De-escalated radiation therapy for patients undergoing surgery to the primary site followed by chemoradiation to the primary site and neck for oropharyngeal squamous cell carcinoma
  Interventions: Radiation: De-escalation

INTERVENTIONS:
Radiation: De-escalation — Surgical resection of primary oropharyngeal tumour followed by de-escalated radiation therapy (30Gy) with concurrent platinum-based chemotherapy to oropharynx + neck, followed by surgical neck dissection
  Arms: De-escalation
Radiation: Standard of care — Radiation therapy (70Gy) with concurrent platinum-based chemotherapy to oropharynx + neck
  Arms: Standard of care

SUMMARY:
The goal of this prospective clinical trial is to determine if HPV-associated oropharyngeal squamous cell carcinoma that is non-hypoxic on FMISO PET can be successfully treated with a lower dose of radiation therapy.

The main questions it aims to answer are:

1. What is the pathologic complete response rate in patients selected for radiation dose de-escalation and neck dissection?
2. What is the correlation between MRI and FMISO PET assessment of hypoxia before and during RT?
3. What are the acute and late toxicities in patients selected for radiation dose de-escalation?
4. What are the quality of life scores in patients selected for radiation dose de-escalation?
5. What are the local, regional and distant failure rates of patients selected for radiation dose de-escalation?

Patients with cT1-2N1-2b (AJCC 7th edition) oropharyngeal tumours will undergo surgical resection of the primary tumour. Following this, they will be allocated to standard radiation therapy (70Gy with concurrent cisplatin chemotherapy) or de-escalation radiation therapy (30Gy with concurrent cisplatin chemotherapy) based on the results of FMISO PET. Patients with non-hypoxic tumours at baseline OR after two weeks of radiation therapy will be allocated to the de-escalated group. 3-4 months after completion of radiation therapy, all patients in the de-escalated group will undergo mandatory neck dissection to assess pathologic response.

Researchers will assess the pathologic response rate after surgery in the de-escalation group. They will also compare the outcomes (oncological outcomes and quality of life) between the group receiving the standard treatment (70Gy) and the group receiving de-escalated radiation therapy (30Gy).

DETAILED DESCRIPTION:
This study is designed to evaluate the role of FMISO PET in selecting patients for de-escalated RT. Patients with cT1-2N-1-2b HPV+ OPC or cTxN1-2 CUP, who are suitable for surgical management of the primary (if applicable) and/or RT to the primary and ipsilateral neck will be included. All patients will undergo surgical resection or core biopsy of the primary site if applicable (negative margins and robotic surgery not mandated) or EUA and tonsillectomy (CUP) and FNA or core biopsy of the cervical lymph node (all patients). Patients will be eligible for inclusion if histopathology is consistent with HPV-associated squamous cell carcinoma or CUP, with p16 positivity (IHC) and HPV positivity (PCR).

Patients enrolled will undergo FMISO PET/CT (after surgery to the primary or EUA/biopsy of suspected primary site) to assess for tumour hypoxia, which will stratify patients into two groups. Determination for the presence or absence of hypoxia will be made on the basis of visual inspection and in accordance with well-established tumour-muscle activity ratio (>1.2) on the late static 18F-FMISO PET by 1 nuclear medicine physician. FMISO PET will be repeat after 5-10 fractions of RT (1-2 weeks of treatment) with the same assessment for hypoxia.

Absence of pre-treatment hypoxia or intra-treatment resolution of hypoxia on FMISO PET will be deemed as an indicator of radiosensitivity and qualify a patient for de-escalation (i.e., to total dose 30Gy). The remainder of patients (i.e., with evidence of tumour hypoxia at the FMISO PET performed after 5-10 fractions of RT) will continue to standard of care RT to a total dose of 70Gy.

Additional MRI images (including T1, T2 and dynamic contract-enhanced and oxygen enhanced sequences) before and during RT (at the same time as 18F FMISO PET). These will not change the patient's management.

All patients will undergo routine FDG-PET/CT scan three months after RT (as part of standard of care). Patients in the de-escalation arm will undergo mandatory ipsilateral neck dissection within 3-4 months of completing RT to assess for pathologic response. Patients will be followed up for a minimum of five years post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically confirmed cT1-2N1-2b oropharyngeal squamous cell carcinoma or cTxN1-2 carcinoma of unknown primary
* p16 positive (70% nuclear and cytoplasmic staining) and HPV positive (genotyping via PCR) tumours of the tonsil, base of tongue, glossotonsillar sulcus, or unknown primary site (suspected mucosal origin).
* No contraindications to radiotherapy, platinum-based chemotherapy or surgery
* No contraindications to PET/CT or MRI
* Eastern Cooperative Oncology Group (ECOG) performance status score 0-2 (KPS > 70%)
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Women lactating, pregnant or of childbearing potential who are not willing to avoid pregnancy during the study
* Patients with a history of severe renal disease(s) (eGFR <20) than cannot tolerate gadolinium chelate contrast agents.)
* ECOG ≥ 3
* Previous high dose radiation therapy to the head or neck
* Patients unwilling or unable to have PET/CT or MRI
* Geographically remote patients unable to agree to imaging schedule
* Patients with a history of psychological illness or condition such as to interfere with the patient's ability to understand the requirements of the study.
* Patients with significant cardiac or pulmonary disease including cardiac arrythmias or Chronic Obstructive Pulmonary Disease (COPD) that are unable to tolerate high flow O2 for oxygen contrast.
* Patients taking carbonic anhydrase inhibitors (acetazolamide)
* History of glaucoma
* Any implant, foreign body, 3T MRI incompatible device, or other contraindication to MRI imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | 4 months after completion of radiation therapy
  Pathologic complete response in surgical neck dissection

SECONDARY OUTCOMES:
Correlation between MRI and FMISO PET assessment of hypoxia | Baseline and after 2 weeks of radiation therapy
  Correlation between MRI and FMISO PET assessment of hypoxia at baseline and during radiation therapy
Quality of Life of patients undergoing de-escalation radiation therapy | Baseline, then 3 months post completion of treatment, then 3-monthly post to 2 years, then 6-monthly to 5 years
  Quality of Life - Global (assessment by EORTC QLQ-30)
Quality of Life of patients undergoing de-escalation radiation therapy | Baseline, then 3 months post completion of treatment, then 3-monthly post to 2 years, then 6-monthly to 5 years
  Quality of Life - Head & Neck Specific (assessment by EORTC HN-35)
Local control | 3-monthly to 2 years, 6-monthly to 5 years
  Failure rate at primary site (oropharynx) (calculated from date of commencing RT)
Regional control | 3-monthly to 2 years, 6-monthly to 5 years
  Failure rate in neck (calculated from date of commencing RT)
Distant metastases | 3-monthly to 2 years, 6-monthly to 5 years
  Number of participants with radiologically confirmed distant metastases (calculated from date of commencing RT)
Acute toxicities | From date of commencement of RT, measured weekly during RT, fortnightly post treatment (up to 3 months post treatment)
  Acute toxicities of radiation therapy +/- chemotherapy (assessed by CTCAE V 5.0)
Late toxicities | Commencing from 3 months post treatment and measured 3-monthly to 2 years, then 6-monthly to 5 years
  Acute toxicities of radiation therapy +/- chemotherapy (assessed by CTCAE V 5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Lawless, Principal Investigator — Royal North Shore Hospital; Sarah Bergamin, Principal Investigator — Royal North Shore Hospital
Locations (1):
- Northern Sydney Cancer Centre, Royal North Shore Hospital, Saint Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No